CLINICAL TRIAL: NCT00145028
Title: Determination of Carboplatin's Optimal Plasmatic Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Dr Laurence GLADIEFF, Institut Claudius Regaud
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 04 GENE 05
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Neoplasms
Keywords: Neoplasms; Carboplatin; optimal exposure; AUC
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Carboplatin

SUMMARY:
To determine Carboplatin's optimal exposures(optimal AUCs)and parameters they depend on.

ELIGIBILITY:
Inclusion Criteria:

* Carcinoma histologically proved and which must be treated by Carboplatin, excepted weekly administered Carboplatin treatments
* Age > 18 years
* Neutrophils > 1500/mm3, blood-platelets > 100000/mm3
* Patient with intravenous administration route for chemotherapy independent of the one used for blood samples ( for Investigators centers achieving pharmacokinetic examination)
* Well-informed written consent, signed by the patient

Exclusion Criteria:

* Carboplatin treatment's contra-indication
* Patient with clinically detectable cerebral metastasis
* Pregnant or nursing women
* Patient under guardianship or trusteeship
* Patient whose venous status don't permit a peripheral intravenous administration route's placing (for Investigators centers achieving pharmacokinetic examination)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine Carboplatin's optimal exposures (optimal AUCs) and parameters they depend on.

SECONDARY OUTCOMES:
To assign a standardization method for Carboplatin doses's calculation in chemotherapy's protocol including this drug.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence GLADIEFF, Doctor, Principal Investigator — Institut Claudius Regaud
Locations (15):
- France (15):
  - Centre Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Clinique Pasteur, Évreux
  - CHU A. Michallon, Grenoble
  - Centre Oscar Lambert, Lille
  - CHU de la Timone, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Hopital Européen Georges Pompidou, Paris
  - Clinique Mathilde, Rouen
  - Centre René Gauducheau, Saint Herblain (Nantes)
  - CHU de Toulouse Rangueil, Toulouse
  - Institut Claudius Regaud, Toulouse
  - CHRU Bretonneau, Tours